CLINICAL TRIAL: NCT01285557
Title: An Open-Label, Multicenter, Randomized, Phase 3 Study of S-1 and Cisplatin Compared With 5-FU and Cisplatin in Patients With Metastatic Diffuse Gastric Cancer Previously Untreated With Chemotherapy
Brief Title: Diffuse Gastric and Esophagogastric Junction Cancer S-1 Trial
Acronym: DIGEST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to significant changes in investigational and clinical practice landscape of frontline advanced gastric cancer, which challenged viability of trial and increased use of modified chemotherapeutic triplets led to slow participant accrual in study.
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPU-S1303
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Results first posted 2022-05-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Diffuse Gastric Cancer Including Carcinoma of the Gastro-esophageal Junction
Keywords: Gastric Cancer , S-1, Phase 3
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); tegafur-gimeracil-oteracil; Cisplatin; titanium silicide; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S-1+Cisplatin (Experimental): Participants received S-1 25 milligrams per meter square (mg/m^2) orally twice daily (BID) every 12 hours from Day 1 through Day 21, 1 hour before or after meal with a glass of water; followed by a 7-day rest period from Day 22 to Day 28 in a 28-day cycle. Participants received a single dose of cisplatin 75 mg/m^2 as a 1- to 3-hour intravenous (IV) infusion on Day 1 following the morning dose of S-1 for a maximum of 8 cycles (each cycle of 28 days). Participants received study medication until progression of disease (PD), adverse event (AE), withdrawal of consent, or other reason for discontinuation, whichever happened earlier.
  Interventions: Drug: S-1 (Tegafur+Gimeracil+Oteracil) /cisplatin (investigational arm)
- 5FU+Cisplatin (Active Comparator): Participants received 5-Fluorouracil (5-FU) 800 mg/m^2 per 24 hours as continuous IV infusion over 120 hours from Day 1 through Day 5 followed by a 16-day rest period on Days 6 through 21 in a 21-day cycle. Participants received a single dose of cisplatin 80 mg/m^2 as a 1- to 3-hour IV infusion on Day 1 prior to the start of the 5-FU infusion on Day 1 for a maximum of 8 cycles (each cycle of 21 days). Participants received study medication until PD, AE, withdrawal of consent, or other reason for discontinuation, whichever happened earlier.
  Interventions: Drug: Fluorouracil/cisplatin (control arm)

INTERVENTIONS:
Drug: S-1 (Tegafur+Gimeracil+Oteracil) /cisplatin (investigational arm) — 25 mg/m² body surface area (BSA) orally 2 times daily from Days 1 through 21 followed by a 7 day rest period, plus cisplatin 75 mg/m2 BSA on Day 1 each 28 day cycle Number of Cycles: until progression or unacceptable toxicity develops. Treatment with cisplatin is limited to a maximum of 8 cycles.
  Other Names: TS-1, Tegafur+Gimeracil+Oteracil
  Arms: S-1+Cisplatin
Drug: Fluorouracil/cisplatin (control arm) — 5-FU: 800 mg/m2 BSA/24 hours by continuous intravenous infusion (CIV) from Days 1 through 5 plus cisplatin 80 mg/m2 BSA on Day 1 each 21 day cycle.
  Number of Cycles: until progression or unacceptable toxicity develops. Treatment with cisplatin is limited to a maximum of 8 cycles.
  Other Names: TS-1, Tegafur+Gimeracil+Oteracil
  Arms: 5FU+Cisplatin

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of S-1 and Cisplatin compared to 5-FU and Cisplatin in treatment of patients with metastatic diffuse gastric and gastro-esophageal junction cancer previously untreated with chemotherapy.

DETAILED DESCRIPTION:
This is an open-label, international, Phase 3 study evaluating the efficacy and safety of the S-1/cisplatin regimen versus the 5-FU/cisplatin regimen in chemotherapy-naïve patients with metastatic diffuse gastric carcinoma including carcinoma of the gastro-esophageal junction. Patients will be randomly assigned to S-1/cisplatin (experimental regimen, Arm A) or 5-FU/cisplatin (control regimen, Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Has given written Informed Consent.
* Histologically confirmed, unresectable, metastatic diffuse gastric cancer including carcinoma of the gastro-esophageal junction.
* No prior chemotherapy for gastric cancer except adjuvant and/or neo-adjuvant chemotherapy more than 12 months ago.
* Life expectancy of at least 3 months.
* Able to take medications orally.
* Eastern Cooperative Oncology Group performance status 0 to 1.
* Adequate organ function (bone marrow, kidney and liver).

Exclusion Criteria:

* Certain type(s) of non-measurable lesion(s), if the only one(s).
* Certain serious illness or medical condition(s).
* Lost greater than or equal to 10% of body weight in the 3 months proceeding signing the Informed Consent Form.
* Treatment with drugs interacting with S-1, 5-FU, or cisplatin.
* Pregnant or lactating female.
* Known hypersensitivity to fluoropyrimidines or cisplatin.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2011-04-14 (Actual); Primary Completion 2014-08-15 (Actual); Study Completion 2014-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Central, Study Director — Taiho Oncology, Inc. USA
Locations (76):
- United States (4):
  - Alexandria, Louisiana
  - Albuquerque, New Mexico
  - Dallas, Texas
  - Houston, Texas
- Argentina (2):
  - Rosario, Santa Fe Province
  - Buenos Aires
- Belgium (3):
  - Brussels
  - Edegem
  - Ghent
- Brazil (9):
  - Salvador, Estado de Bahia
  - Porto Alegre, Rio Grande do Sul
  - Barretos, São Paulo
  - Ribeirão Preto, São Paulo
  - São Paulo, São Paulo
  - Belo Horizonte
  - Fortaleza
  - Ijuí
  - Porto Alegre
- Bulgaria (2):
  - Pleven
  - Vratsa
- Croatia (2):
  - Osijek
  - Zagreb
- Tallinn, Estonia
- Essen, Germany
- Hungary (6):
  - Budapest
  - Győor
  - Nyíregyháza
  - Pécs
  - Szeged
  - Székesfehérvár
- Tel Aviv, Israel
- Italy (7):
  - Ancona
  - Candiolo
  - Milan
  - Modena
  - Potenza
  - Reggio Emilia
  - Rimini
- Mexico (3):
  - Chihuahua City
  - Mexico City
  - Oaxaca City
- Poland (2):
  - Szczecin
  - Warsaw
- Portugal (4):
  - Aveiro
  - Coimbra
  - Lisbon
  - Porto
- Romania (4):
  - Baia Mare
  - Cluj-Napoca
  - Craiova
  - Iași
- Russia (5):
  - Barnaul
  - Krasnodar
  - Moscow
  - Pyatigorsk
  - Saint Petersburg
- South Africa (4):
  - Groenkloof Pretoria, Gauteng
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Cape Town, Western Cape
- Spain (3):
  - Sabadell, Barcelona
  - Barcelona
  - Madrid
- Ukraine (11):
  - Cherkassy
  - Chernivtsiy
  - Dnipro
  - Donetsk
  - Kharkiv
  - Kyiv
  - Lutsk
  - Lviv
  - Sumy
  - Uzhhorod
  - Zaporizzhya
- United Kingdom (2):
  - Rhyl, Wales
  - London

REFERENCES:
- [Derived] Ajani JA, Abramov M, Bondarenko I, Shparyk Y, Gorbunova V, Hontsa A, Otchenash N, Alsina M, Lazarev S, Feliu J, Elme A, Esko V, Abdalla K, Verma U, Benedetti F, Aoyama T, Mizuguchi H, Makris L, Rosati G; DIGEST Study Group. A phase III trial comparing oral S-1/cisplatin and intravenous 5-fluorouracil/cisplatin in patients with untreated diffuse gastric cancer. Ann Oncol. 2017 Sep 1;28(9):2142-2148. doi: 10.1093/annonc/mdx275. PMID 28911091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 690 participants were screened from 14 April 2011 to 25 February 2014, of which 361 participants enrolled in the study. The data cut-off date for all clinical data except overall survival was 07 Mar 2014 and for overall survival was 15 Aug 2014. The participants were randomized using interactive Voice/Web randomization system(2:1 ratio) to receive S-1/cisplatin or 5-Fluorouracil (5-FU)/cisplatin. A total of 329 participants failed screening due to failure to meet inclusion criteria.
Pre-assignment Details: Randomization was stratified by the histologic subtype (adenocarcinoma, diffuse type or signet ring cell adenocarcinoma); extent of metastasis (1 versus more than 1 metastatic site); Eastern Cooperative Oncology Group (ECOG) performance status (0 or 1) and region (North America, Western Europe, Eastern Europe, Rest of world). Cut-off dates for all clinical data collection was 07 March 2014 and for overall survival analysis was 15 August 2014.
Groups:
- 5FU+Cisplatin: Participants received 5-FU 800 mg/m^2 per 24 hours as continuous IV infusion over 120 hours from Day 1 through Day 5 followed by a 16-day rest period on Days 6 through 21 in a 21-day cycle. Participants received a single dose of cisplatin 80 mg/m^2 as a 1- to 3-hour IV infusion on Day 1 prior to the start of the 5-FU infusion on Day 1 for a maximum of 8 cycles (each cycle of 21 days). Participants received study medication until PD, AE, withdrawal of consent, or other reason for discontinuation, whichever happened earlier.
Period: Overall Study
Arm/Group | S-1+Cisplatin | 5FU+Cisplatin
Started | 239 | 122
Treated | 238 | 121
As Treated (AT) Population (Participants started either of 2 treatment regimens assigned according to actual treatment received.) | 230 | 118
Completed | 0 | 0
Not Completed | 239 | 122
Not completed — Death | 173 | 90
Not completed — Lost to Follow-up | 6 | 2
Not completed — Withdrew Consent | 6 | 1
Not completed — Sponsor Study Termination | 23 | 13
Not completed — Randomized but not treated | 1 | 1
Not completed — Study follow-up ongoing | 28 | 14
Not completed — Sponsor Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all randomized participants including those not dosed according to their randomization.
Groups:
- S-1+Cisplatin: Participants received S-1 25 mg/m^2 orally BID every 12 hours from Day 1 through Day 21, 1 hour before or after meal with a glass of water; followed by a 7-day rest period from Day 22 to Day 28 in a 28-day cycle. Participants received a single dose of cisplatin 75 mg/m^2 as a 1- to 3-hour IV infusion on Day 1 following the morning dose of S-1 for a maximum of 8 cycles (each cycle of 28 days). Participants received study medication until PD, AE, withdrawal of consent, or other reason for discontinuation, whichever happened earlier.
- Total: Total of all reporting groups
Arm/Group | S-1+Cisplatin | 5FU+Cisplatin | Total
Number analyzed (Participants) | 239 | 122 | 361
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (11.01) | 55.8 (11.80) | 55.4 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 62 | 177
  Male | 124 | 60 | 184
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 226 | 117 | 343
  Black | 4 | 2 | 6
  Asian/Oriental | 4 | 0 | 4
  American Indian or Alaska Native | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 3 | 3 | 6
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG performance status was used to evaluate participant's disease progression and the effect of the disease on the participant's activities of daily living. It ranged on the scale from 0-5 (0 equal to [=] normal activity; 1= symptoms but ambulatory; 2= in bed for less than (<) 50 percent (%) of the time; 3= in bed for greater than (>) 50% of the time; 4= 100% bedridden; 5= dead).
  Participants
    ECOG Grade 0 | 75 | 38 | 113
    ECOG Grade 1 | 164 | 83 | 247
    Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death for the ITT population. Participants who did not die were censored at the date last known to be alive. Analysis was performed by using Kaplan-Meier method.
Time Frame: From the date of randomization until disease progression or death, cut-off date: 15 August 2014 (approximately 40 months)
Population: Analysis was performed on the ITT population that included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | S-1+Cisplatin | 5FU+Cisplatin
Number analyzed (Participants) | 239 | 122
months | 7.5 [6.7 to 9.3] | 6.6 [5.7 to 8.1]
Statistical Analysis 1: Comparison: S-1+Cisplatin vs 5FU+Cisplatin; S-1+Cisplatin and 5FU+Cisplatin were compared using the unstratified log-rank test. The hazard ratio was estimated using a Cox's regression approach and survival was summarized using Kaplan Meier estimates along with 2-sided 95% confidence intervals (CI) for the estimates; Test type: Superiority; p = 0.9312, Unstratified Log-rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.76 to 1.28]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from date of randomization until date of radiological disease progression or death due to any cause. Disease Progression was defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, where any of the 3 criteria have been met: 1) at least 20% increase in the sum of diameters of the target lesions, taking as reference the smallest sum on study, including the baseline sum, 2) Progression in no-target lesion(s), 3) appearance of new lesion(s) Participants who were alive with no PD were censored at the date of the last tumor assessment. Participants who received new anticancer therapy before disease progression were censored at the date of the last evaluable tumor assessment before new anticancer therapy was initiated. Analysis was performed by using Kaplan-Meier method.
Time Frame: From date of randomization until disease progression or death, cut-off date: 07 March 2014 (approximately 34.7 months)
Population: Analysis was performed on the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | S-1+Cisplatin | 5FU+Cisplatin
Number analyzed (Participants) | 239 | 122
months | 4.4 [3.8 to 5.6] | 3.9 [3.6 to 5.2]
Statistical Analysis 1: Comparison: S-1+Cisplatin vs 5FU+Cisplatin; S-1+Cisplatin and 5FU+Cisplatin were compared using the log-rank test. The hazard ratio was estimated using a Cox's regression approach and survival was summarized using Kaplan Meier estimates along with 2-sided 95% confidence intervals (CI) for the estimates; Test type: Superiority; p = 0.3039, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.65 to 1.14]

3. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF was defined as the time from date of randomization until date of PD (clinical or radiologic), or permanent discontinuation of study treatment (S-1 or 5-FU), or death due to any cause. Participates who were still on study treatment at the time of the analysis were censored at the last date the participants was known to be on treatment.
Time Frame: From date of randomization until disease progression, cut-off date: 07 March 2014 (approximately 34.7 months)
Population: Analysis was performed on the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | S-1+Cisplatin | 5FU+Cisplatin
Number analyzed (Participants) | 239 | 122
months | 4.2 [3.8 to 4.9] | 3.8 [3.4 to 4.3]
Statistical Analysis 1: Comparison: S-1+Cisplatin vs 5FU+Cisplatin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1683, Log Rank; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.66 to 1.08]

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAE)
Description: AE was defined as any untoward medical condition that occurs in a participants while participating in a clinical study and does not necessarily had to have a causal relationship with the use of the study medication. A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs were defined as AEs that developed or worsened or became serious during on-treatment period (from first dose of study medication up to 30 days of last study medication [maximum duration: 35.7 months]).
Time Frame: From first dose of study medication up to 30 days of last study medication (maximum duration: 35.7 months)
Population: Analysis was performed on the as treated (AT) population that included all participants who initiated treatment with either of the 2 regimens with treatment assignment designated according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | S-1+Cisplatin | 5FU+Cisplatin
Number analyzed (Participants) | 230 | 118
Participants
  TEAE | 214 | 111
  TESAE | 63 | 31

5. Secondary Outcome: Number of Participants With TEAEs With Severity Greater Than or Equal to (>=) Grade 3
Description: An AE was any untoward medical condition that occurred in a participants while participating in a clinical study and does not necessarily had to have a causal relationship with the use of the study medication. TEAEs were defined as AEs that developed or worsened or became serious during on-treatment period (from first dose of study medication up to 30 days of last study medication [maximum duration: 35.7 months]).
Time Frame: From first dose of study medication up to 30 days of last study medication (maximum duration: 35.7 months)
Population: Analysis was performed on the as treated (AT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | S-1+Cisplatin | 5FU+Cisplatin
Number analyzed (Participants) | 230 | 118
Participants | 157 | 78

6. Secondary Outcome: Overall Response Rate (ORR): Percentage of Participants With Overall Response
Description: ORR was defined as the percentage of participants with objective evidence of complete response (CR) or partial response (PR) based on the Investigator review of the images and application of Response Evaluation Criteria in Solid Tumors (RECIST) criteria. CR was defined as the disappearance of all target or non-target lesions. Any pathological lymph nodes for target lesions or all lymph nodes for non-target lesions were non-pathological morphologically that was reduced in size in short axis to less than (<) 10 millimeter (mm). PR was defined as target lesions with at least 30% decrease in the sum of diameters, taking baseline sum diameters as reference.
Time Frame: From date of first study medication until cut-off date: 07 March 2014 (approximately 34.7 months)
Population: Analysis was performed on the ITT population. Here, 'overall number of participants analyzed' signifies participants with available data for the outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | S-1+Cisplatin | 5FU+Cisplatin
Number analyzed (Participants) | 193 | 91
percentage of participants | 34.7 [28.0 to 41.9] | 19.8 [12.2 to 29.4]

7. Secondary Outcome: Duration of Response (DR)
Description: Duration of response was defined as the time (in months) from date of first confirmed response (CR or PR) to date of first progressive disease (PD) or death. Per the RECIST criteria, definitions were as follows: CR was defined as the disappearance of all target or non-target lesions. Any pathological lymph nodes for target lesions or all lymph nodes for non-target lesions were non-pathological morphologically that was reduced in size in short axis to <10 mm. Analysis was performed by using Kaplan-Meier method.
Time Frame: From date of first study medication until cut-off date: 07 March 2014 (approximately 34.7 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | S-1+Cisplatin | 5FU+Cisplatin
Number analyzed (Participants) | 67 | 18
months | 5.1 [3.0 to 5.8] | 4.2 [2.0 to 6.0]

8. Secondary Outcome: Time to Tumor Response (TTR)
Description: TTR was defined as the time (in months) from the date of randomization to the date of first observation of response (PR or CR) (whichever status was recorded first). TTR was assessed based on investigator assessment utilizing RECIST 1.1. CR was defined as the disappearance of all target or non-target lesions. Any pathological lymph nodes for target lesions or all lymph nodes for non-target lesions were non-pathological morphologically that was reduced in size in short axis to <10 mm. PR was defined as target lesions with at least 30% decrease in the sum of diameters, taking baseline sum diameters as reference. Analysis was performed by using Kaplan-Meier method.
Time Frame: From date of first study medication until cut-off date: 07 March 2014 (approximately 34.7 months)
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | S-1+Cisplatin | 5FU+Cisplatin
Number analyzed (Participants) | 67 | 18
months | 1.8 [1.8 to 1.9] | 1.9 [1.8 to 2.1]

ADVERSE EVENTS:
Time Frame: AEs were collected from first dose of study medication up to 30 days of last study medication (maximum duration: 35.7 months). Deaths were collected from Baseline up to end of study (up to approximately 40 months).
Description: Reported AEs were TEAEs. TEAEs were defined as AEs that developed or worsened or became serious during on-treatment period (defined as the time from first dose of study medication up to 30 days of last study medication) and was assessed on AT population. All-Cause Mortality data collected during the study was assessed on all randomized participants.
Arm/Group | S-1+Cisplatin | 5FU+Cisplatin
All-Cause Mortality (participants affected / at risk) | 173/239 | 90/122
Serious Adverse Events (participants affected / at risk) | 63/230 | 31/118
Other Adverse Events (participants affected / at risk) | 210/230 | 110/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-1+Cisplatin (N=230) | 5FU+Cisplatin (N=118)
Anaemia (Blood and lymphatic system disorders) | 11 (12) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cytotoxic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 3 (3) | 4 (4)
Gastric perforation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (5) | 2 (3)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (4)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 1 (1)
Device occlusion (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 5 (5) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S-1+Cisplatin (N=230) | 5FU+Cisplatin (N=118)
Anaemia (Blood and lymphatic system disorders) | 97 (160) | 49 (86)
Granulocytopenia (Blood and lymphatic system disorders) | 13 (59) | 5 (8)
Leukopenia (Blood and lymphatic system disorders) | 31 (80) | 12 (23)
Neutropenia (Blood and lymphatic system disorders) | 68 (161) | 43 (92)
Thrombocytopenia (Blood and lymphatic system disorders) | 37 (74) | 10 (12)
Tinnitus (Ear and labyrinth disorders) | 19 (27) | 11 (22)
Abdominal distension (Gastrointestinal disorders) | 18 (33) | 5 (11)
Abdominal pain (Gastrointestinal disorders) | 42 (62) | 12 (14)
Abdominal pain upper (Gastrointestinal disorders) | 16 (20) | 10 (10)
Ascites (Gastrointestinal disorders) | 13 (15) | 8 (8)
Constipation (Gastrointestinal disorders) | 39 (52) | 17 (32)
Diarrhoea (Gastrointestinal disorders) | 41 (74) | 22 (46)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 6 (8) | 8 (13)
Nausea (Gastrointestinal disorders) | 122 (272) | 62 (131)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 18 (36)
Vomiting (Gastrointestinal disorders) | 82 (142) | 34 (59)
Asthenia (General disorders) | 55 (80) | 36 (61)
Fatigue (General disorders) | 59 (104) | 28 (51)
Mucosal inflammation (General disorders) | 20 (23) | 19 (36)
Oedema peripheral (General disorders) | 17 (20) | 7 (9)
Pyrexia (General disorders) | 19 (27) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 12 (13) | 4 (4)
Blood bilirubin increased (Investigations) | 13 (17) | 1 (1)
Blood creatinine increased (Investigations) | 20 (26) | 8 (11)
Creatinine renal clearance decreased (Investigations) | 9 (9) | 8 (10)
Weight decreased (Investigations) | 40 (42) | 18 (18)
Decreased appetite (Metabolism and nutrition disorders) | 95 (184) | 40 (68)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 7 (13)
Hypomagnesaemia (Metabolism and nutrition disorders) | 24 (30) | 9 (11)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (7) | 6 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 5 (7)
Headache (Nervous system disorders) | 18 (32) | 7 (7)
Neuropathy peripheral (Nervous system disorders) | 23 (28) | 14 (17)
Insomnia (Psychiatric disorders) | 13 (14) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (26) | 8 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 13 (16) | 6 (8)
Dizziness (Vascular disorders) | 15 (32) | 1 (1)

LIMITATIONS AND CAVEATS:
Enrollment closure and study termination was due to significant changes in investigational and clinical practice landscape of frontline advanced gastric cancer, which challenged viability of trial and increased use of modified chemotherapeutic triplets led to slow participant accrual in the study. The decision to halt further accrual was not based on any safety or study quality concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes